CLINICAL TRIAL: NCT02867605
Title: Human Pilot Study - HA35 (Hyaluronan Molecular Weight 35) Dietary Supplement for Promoting Intestinal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Carol De La Motte, Assoiciate Staff, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-142
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Gastrointestinal Microbiome
MeSH Terms: interventions — Hyaluronic Acid

ARMS (1):
- Healthy Controls ages 18-45 with BMI of 19-25 or 30-35 (Other): Single Arm study
  Interventions: Dietary Supplement: Hyaluronan

INTERVENTIONS:
Dietary Supplement: Hyaluronan

SUMMARY:
The purpose of this study is to evaluate whether oral HA35 supplementation changes the normal intestinal bacteria, increases intestinal protection, decrease intestinal inflammation and permeability, and to assess any health benefits and confirm the safety profile of HA35.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-25 (lean), and BMI 30-35 (obese)
* Age 18-45 years old
* Willingness to take oral supplement and adhere to study requirements

Exclusion Criteria:

* Diabetes
* Oral antibiotics within 4 weeks of study initiation
* History of cardiac disease, and medications for cardiac disease
* Use statins and antihypertensive drugs
* Inflammatory bowel disease including irritable bowel syndrome
* History of intestinal surgery, excluding hernia repair and appendectomy
* Active cancer diagnosis (except skin cancer)
* Chronic acid suppression treatment (proton pump inhibitors, histamine H2 receptor antagonists)
* Immune modulatory treatments (e.g. chronic immunosuppressive medications, chronic NSAIDs)
* Vegetarian or vegan diet7
* Abnormal liver or kidney function as measured by routine serum chemistry testing
* Severe anemia or significant white blood cell or platelet abnormalities
* No additional blood or blood product donations during the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Hill DR, Kessler SP, Rho HK, Cowman MK, de la Motte CA. Specific-sized hyaluronan fragments promote expression of human beta-defensin 2 in intestinal epithelium. J Biol Chem. 2012 Aug 31;287(36):30610-24. doi: 10.1074/jbc.M112.356238. Epub 2012 Jul 3. PMID 22761444
- [Background] Hill DR, Rho HK, Kessler SP, Amin R, Homer CR, McDonald C, Cowman MK, de la Motte CA. Human milk hyaluronan enhances innate defense of the intestinal epithelium. J Biol Chem. 2013 Oct 4;288(40):29090-104. doi: 10.1074/jbc.M113.468629. Epub 2013 Aug 15. PMID 23950179

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls Ages 18-45 With BMI of 19-25 or 30-35: Hyaluronan
Period: Overall Study
Arm/Group | Healthy Controls Ages 18-45 With BMI of 19-25 or 30-35
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Controls Ages 18-45 With BMI of 19-25 or 30-35
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Composition of Stool Micro Biome Diversity and Phylogenetic Distribution at 0 Days, 8 Days and 28 Days
Description: Relative abundance is defined as the proportion of total identified bacteria in a sample that are a given type of bacteria. As an example a relative abundance of firmicutes equal to 0.9 would mean that 90% of the bacteria identified in a sample are firmicutes
Time Frame: Baseline, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Day 0: Baseline/Pre Treatment
- Day 8: Immediately post 7 day treatment
- Day 28: 28 days post treatment
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
ratio
  firmicutes | 0.697 (0.164) | 0.722 (0.133) | 0.735 (0.118)
  actinobacteria | 0.146 (0.0985) | 0.145 (0.111) | 0.141 (0.0951)
  bacteroidetes | 0.0969 (0.0855) | 0.00789 (0.0497) | 0.101 (0.102)
  verrucomicrobia | 0.0415 (0.117) | 0.0398 (0.115) | 0.0151 (0.0273)
  proteobacteria | 0.0111 (0.0211) | 0.00789 (0.0118) | 0.00432 (0.00509)
  euryarchaeota | 0.00381 (0.00797) | 0.00295 (0.00558) | 0.00221 (0.00463)
  tenericutes | 0.00275 (0.00605) | 0.00267 (0.00602) | 0.00152 (0.00322)
  unclassified | 0.000272 (0.00000633) | 0.000243 (0.00000618) | 0.000237 (0.00000733)
  others | 0.000359 (0.000589) | 0.000134 (0.000247) | 0.000183 (0.00031)

2. Primary Outcome: Laboratory Parameters at Day 0, Day 8 and 28 Calcium, Bilirubin, Glucose, Blood Urea Nitrogen, Creatinine
Time Frame: Baseline, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Day 8: Immediately post 7 days of treatment
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
mg/dL
  Calcium | 9.2 (0.4) | 9.2 (0.2) | 9.1 (0.3)
  Bilirubin (total) | 0.4 (0.3) | 0.4 (0.2) | 0.4 (0.3)
  Glucose | 92 (20) | 94 (16) | 89 (27)
  blood urea nitrogen | 11 (3) | 11 (4) | 12 (3)
  Creatinine | 0.85 (0.16) | 0.85 (0.16) | 0.83 (0.15)

3. Primary Outcome: Indirect Calorimetry Data at 0 Day, 8 Days and 28 Days Volume of Oxygen and Volume Carbon Dioxide
Time Frame: Baseline, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Day 0: Baseline/ Pretreatment
- Day 8: immediately post treatment
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
L/min
  volume oxygen | 0.225 (0.041) | 0.224 (0.039) | 0.239 (0.048)
  volume carbon dioxide | 0.180 (0.029) | 0.184 (0.035) | 0.197 (0.038)

4. Primary Outcome: Indirect Calorimetry Data at 0 Day, 8 Days and 28 Days Respiratory Quotient RQ
Description: The respiratory quotient is a ratio between the volume of carbon dioxide exhaled and the volume of oxygen inhaled during respiration. It typically ranges between 0.7 and 1.0 and is an indicator of metabolic fuel or substrate use in tissues; it must be calculated under resting or steady-state exercise conditions. A ratio of 0.7 is indicative of mixed fat use, whereas a ratio of 1.0 indicates the exclusive use of carbohydrates
Time Frame: Baseline, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Day 0: Baseline/pretreatment
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
ratio | 0.808 (0.077) | 0.822 (0.061) | 0.826 (0.0708)

5. Primary Outcome: Fecal Intestinal Antimicrobial Peptide Secretion at 0 Days, 8 Days and 28 Days Total Protein
Time Frame: Baseline, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
ug/mL | 22883.8 (6425.7) | 22365.3 (5872.8) | 22726.3 (6305.2)

6. Primary Outcome: Fecal Intestinal Antimicrobial Peptide Secretion at 0 Days, 8 Days and 28 Days Normalized Calprotectin and Human Beta-Defensin2
Time Frame: Baseline, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: ng/ug
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
ng/ug
  calprotectin | 0.00627 (0.0033) | 0.00828 (0.005886) | 0.00891 (0.00557)
  human beta-Defensin2 | 0.0042 (0.00660) | 0.00535 (0.01046) | 0.00362 (0.00814)

7. Primary Outcome: Serum Indicators of Intestinal Permeability at 0 Days, 8 Days and 28 Days Serum Lipopolysaccharide, Hyaluronan
Time Frame: Baseline, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
ng/mL
  Lipopolysaccharide | 0.409 (1.347) | 2.677 (5.959) | 1.256 (4.029)
  Hyaluronan | 338.8 (82.8) | 329.0 (106.6) | 338.7 (73.9)

8. Primary Outcome: Serum Indicators of Inflammation and Injury at Baseline, 8 Days and 28 Days-tumor Necrosis Factor (TNF) Alpha, Interleukin 6 (IL-6)
Time Frame: Baseline, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
pg/mL
  TNF alpha | 2.0 (5.1) | 2.4 (6.6) | 3.2 (6.9)
  interleukin 6 (IL-6) | 9.6 (14.6) | 11.7 (16.8) | 10.5 (14.6)

9. Primary Outcome: Baseline Serum Indicators of Inflammation and Injury at Baseline, 8 Days and 28 Days-C-reactive Protein
Time Frame: Baseline, Day 8, Day 28
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Day 0: Baseline/Pre-treatment
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
g/dL | 10.2 (15.5) | 10.3 (12.8) | 11.6 (13.7)

10. Primary Outcome: Blood Protein, Hemoglobin and Albumin Levels at Baseline, Day 8, and Day 28
Time Frame: Baseline, day 8 day 28
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
g/dL
  Hemoglobin | 13.4 (1.5) | 13.4 (1.4) | 13.2 (1.5)
  Protein | 7.4 (0.3) | 7.3 (0.4) | 7.3 (0.4)
  Albumin | 4.4 (0.3) | 4.4 (0.3) | 4.3 (0.3)

11. Primary Outcome: White Blood Cell and Platelet Count at Baseline, Day 8, and Day 28
Time Frame: baseline, day 8, and day 28
Measure: Mean (Standard Deviation); unit: k/uL
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
k/uL
  White Blood Cell | 6.0 (1.6) | 6.1 (1.4) | 6.2 (1.5)
  Platelet Count | 263 (59) | 262 (63) | 271 (64)

12. Primary Outcome: Alkaline Phosphatase, Alanine Transaminase , and Aspartate Transaminase at Baseline, Day 8, and Day 28
Time Frame: baseline, day 8, and day 28
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
U/L
  Alkaline Phosphatase | 66 (16) | 66 (17) | 67 (17)
  aspartate transaminase | 18 (6) | 22 (18) | 19 (7)
  alanine transaminase | 16 (7) | 15 (6) | 18 (17)

13. Primary Outcome: Serum Sodium, Potassium, and Carbon Dioxide at Baseline Day 8 and Day 28
Time Frame: baseline, day 8, and day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
mmol/L
  Sodium | 140 (1) | 140 (2) | 140 (2)
  Potassium | 4.0 (0.2) | 4.1 (0.3) | 4.0 (0.2)
  carbon dioxide | 25 (2) | 24 (2) | 24 (2)

14. Primary Outcome: Resting Energy Expenditure (REE) and Metabolic Rate at Baseline Day 8 an Day 28
Time Frame: Baseline, day 8, and day 28
Measure: Mean (Standard Deviation); unit: kilocalories/day
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
kilocalories/day
  Resting Energy Expenditure | 1556.3 (274.5) | 1562.8 (221.4) | 1670.6 (333.9)
  Metabolic Rate | 1653.1 (268.7) | 1665.2 (258.8) | 1668.4 (259.8)

15. Primary Outcome: Resting Energy Expenditure as a Percent of Predicted at Baseline, Day 8, and Day 28
Description: This values measures the amount of energy a person uses during rest and compares it the average expected number of someone who is the same gender, age, and race.
Time Frame: Baseline, day 8, and day 28
Measure: Mean (Standard Deviation); unit: percent of age/gender predicted values
Arm/Group | Day 0 | Day 8 | Day 28
Number analyzed (Participants) | 20 | 20 | 20
percent of age/gender predicted values | 95.89 (9.48) | 95.67 (12.94) | 101.39 (10.41)

ADVERSE EVENTS:
Time Frame: 0-28 days
Arm/Group | Day 0 | Day 8 | Day 28
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT02867605/Prot_SAP_001.pdf